CLINICAL TRIAL: NCT04671992
Title: Ultrasound Guided Out Of-Plane Technique Against İn-Plane Technique for Caudal Block in Pediatric Hypospadias Surgery: A Prospective Randomized Clinical Study
Brief Title: Out Of-plane Technique Against In-plane for Caudal Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, Principal investigator, Selcuk University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: farukcicekci3
Record Dates: First submitted 2020-12-06; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Ultrasound Imaging; Caudal Block; Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Out of-Plane Technique (Active Comparator): Ultrasound Guided Out of plane technique (probe applied by holding horizontal)
  Interventions: Device: Out of-Plane Technique and In-Plane on
- Ultrasound Guided In-Plane Technique (Active Comparator): Ultrasound Guided Out of plane technique (probe applied by holding vbertical)
  Interventions: Device: Out of-Plane Technique and In-Plane on

INTERVENTIONS:
Device: Out of-Plane Technique and In-Plane on — A comparison of out of-plane technique and in-plane

SUMMARY:
Caudal block is an easy and effective type of central neuraxial block that is widely used in subumbilical surgeries to provide intraoperative and postoperative analgesia in the pediatric population. Caudal block application with ultrasound (USG) was first applied in 2003. Sacrum, sacral cornular, sacrococcygeal ligament and sacral hiatus can be easily distinguished by ultrasound. The probe is positioned in a horizontal midline position on the lower sacrum. Sacral roots within the caudal epidural space can be seen as hypoechoic ellipses. In addition, anatomical variations of the sacral hiatus and the process area can be clearly observed. A accurate probe use with ultrasound guided is confirmed by advancing the caudal needle in the desired direction, widening in the sacral hiatus with local anesthetic injection, and the turbulence observed during injection into the sacral canal if the color doppler feature is used. Thus, a decrease in complications and an increase in the success of the procedure can be achieved with simultaneous imaging. In addition, in cases where the block is difficult, the in-plane technique can be preferred in the midline plane.The aim of this study is to compare the success rates and postoperative pain levels of caudal block applications with the out of plane technique (probe applied by holding horizontal) and in-plane technique (probe applied vertically), which is routinely applied with ultrasound in pediatric hypospadias surgery.

DETAILED DESCRIPTION:
This study will be scheduled between January - March 2021 at Selcuk University Department of Anesthesiology and Reanimation. A total of 70 patients from American Society of Anesthesiologists classification physical status of (ASA-PS) I-II, aged 6 months to 10 years, will be included in the study. Routine monitoring electrocardiogram (ECG), peripheral oxygen saturation (SpO2) and non-invasive blood pressure measurements will be made to patients into the operating room, and their basal levels will be recorded. All patients were transferred to the operating room without premedication. The patients will be assigned to two groups as in-plane technique (Group IP) and out of-plane technique (Group OP) according to the program randomization list. Routine anesthesia induction will be performed with 7-8% sevoflurane, 100% oxygen until the patient loses consciousness with a face mask. Then, vascular access will be established and propofol 2-3 mg for general anesthesia induction. kg 1 and fentanyl 1 μg. kg-1 IV will be used. After the eyelash reflex disappears without any neuromuscular blocker medication, a suitable laryngeal mask airway device will be placed into supraglottic area, and the patient will be connected to the anesthesia device for ventilation. For the maintenance of anesthesia, 2% sevoflurane, nitrous oxide will be stopped, and 50% oxygen + air mixture will be used. For caudal epidural block, the patient will be turned to the lateral position. After the asepsis of the perianal region is achieved, the sterile 8-18 MHz lineer USG probe for Group OP will be placed transversely in the midline to obtain a transverse view in the sacral hiatus. For group IP, the probe will be rotated 90 degrees and applied with the in-plane technique. After it is observed that there is no blood or cerebrospinal fluid (CSF) with aspiration, local anesthetic (LA) injection will be performed under hemodynamic and ECG monitoring by calculating the dose as 0.5 mg.kg-1 (0.25% bupivacaine) and the volume as 0.5 ml.kg-1. A successful block will be defined as the absence of significant motor movements after surgical induction, after heart and respiratory rates do not increase up to 20% above basal levels. In addition, block application time, number of needle attempts, success at first entry, ease of visualization, LA spread will be recorded and evaluated as the success rate.

In both groups, the surgical caudal block will begin 10 minutes after anesthesia. Intraoperative opioids or sedative drugs will not be used. Mean arterial pressure, heart rate and oxygen saturation of the patients will be recorded every 5 minutes.

At the end of the surgery, patients will be extubated and followed up in the postoperative recovery unit. Postoperative pain 10 minutes, 30 minutes, 1st, 2nd, 3rd, 6th, 12th, 24th hours FLACC pain scale (Face Legs Activity Cry Consolabity = face , legs, activity, crying, consolation). Time to first analgesia requirement, total analgesic consumption and postoperative complications will be recorded. In the evaluations made to patients in both groups, if the FLACC scale is> 4, rescue analgesia will be administered intravenously with 15 mg.kg-1 paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing hypospadias surgery
* ASA PS I-II group

Exclusion Criteria:

* Previous neurological or spinal disorder,
* Coagulation anomaly
* Allergy to local anesthetics
* Local infection in the block area
* Children with a history of preterm birth

Ages: 6 Months to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
the success rates of in-plane and out of-plane techniques | 4 months
  To measure success rates of in-plane and out-of-plane techniques for caudal block, the number of successful processing and the time of processing (minute) will be used

SECONDARY OUTCOMES:
The postoperative pain levels | 4 months
  Postoperative pain will be evaluated with the visual analog scale (VAS), the first analgesia requirement time will to be shown as "minute" and the total amount of analgesia consumed as "mg".

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, School of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not have a plan to make individual participant data (IPD) available to other researchers.